CLINICAL TRIAL: NCT04374409
Title: A Placebo-controlled, Randomized, Double-masked, Cross-over Acute Intervention Study Investigating the Effects of Flavanols on Cerebral Oxygenation and Cognition in Young Adults
Brief Title: Effects of Acute Intake of Flavanols on Cerebral Oxygenation and Cognition in Young Male Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Catarina Rendeiro, Principal Investigator, University of Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ERN_17_1591
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: flavanol; cocoa; brain; oxygenation; vascular; cognition; hypercapnia; functional near-infrared spectroscopy
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flavanol Cocoa powder (Experimental): Dietary supplement: single serving of a high-flavanol cocoa powder containing 150 mg of (-)-epicatechin and 35.5 mg of (+)-catechin
  Interventions: Dietary Supplement: High-flavanol cocoa powder
- Low-flavanol Cocoa powder (Active Comparator): Dietary supplement: single serving of a low-flavanol cocoa powder intervention containing < 4 mg of (-)-epicatechin and (+)-catechin and matched as best as possible for macronutrients and micronutrients, such as caffeine and theobromine.
  Interventions: Dietary Supplement: Low-flavanol cocoa powder

INTERVENTIONS:
Dietary Supplement: High-flavanol cocoa powder — Non-alkalized fat-reduced cocoa powder (Natural Acticoa)
  Arms: High-flavanol Cocoa powder
Dietary Supplement: Low-flavanol cocoa powder — Alkalized fat-reduced cocoa powder (10/12 DDP Royal Dutch)
  Arms: Low-flavanol Cocoa powder

SUMMARY:
The study evaluates the impact of one acute dose of cocoa flavanols on brain oxygenation during a hypercapnia challenge, as well as impact on cognitive performance in young healthy males. It further assesses the impact of flavanols on peripheral vascular function, as measured by brachial Flow-mediated dilation (FMD). All participants received a high-flavanol cocoa intervention (185.5 mg of flavanols (-)-epicatechin and (+)- catechin) and a low-flavanol cocoa intervention (< 4 mg of flavanols). It is hypothesized that the high-flavanol intervention increases cerebral oxygenation during hypercapnia and vascular function in comparison to the low-flavanol intervention.

DETAILED DESCRIPTION:
Cocoa flavanols have been shown to be protective against vascular disease in humans, as evidenced by improvements in peripheral endothelial function (as measured by brachial Flow-mediated dilatation, FMD). There is also emerging evidence suggesting that flavanol-rich diets protect against cognitive aging, but mechanisms remain elusive. In this study the investigators suggest that such mechanisms might be associated with benefits within the brain vasculature. The aim of the present study was therefore to determine whether intake of flavanols enhances cerebral oxygenation in frontal cortical areas of the brain during a hypercapnia challenge (which is a well-established biomarker of vascular reactivity in the brain) to a greater extent than a low-flavanol intervention in young healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-45 years old

Exclusion Criteria:

* smokers
* hypertensive
* with history of cerebrovascular, cardiovascular or respiratory disease
* allergies or intolerances to ingredients present in cocoa powders
* taking long-term medication (e.g., hyperlipidaemia)
* on antibiotics for the previous 3 months before enrollment
* suffering from blood-clotting disorders
* known infections at the time of the study
* on a weight-reducing regimen

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Cortical Blood Oxygenation reactivity to hypercapnia using functional near-infrared spectroscopy (fNIRS) | Change from baseline to 2 hours
  Cerebral oxygenated haemoglobin maximum levels in the frontal cortical regions of the brain during the 5% carbon-dioxide breathing challenge (average across minutes 3 and 4 of breathing challenge)
Time to reach 90% of maximum cortical blood oxygenation during hypercapnia using functional near-infrared spectroscopy (fNIRS) | Change from baseline to 2 hours
  Time to reach 90% of maximum oxygenated haemoglobin in the frontal cortical regions of the brain during the 5% carbon-dioxide breathing challenge

SECONDARY OUTCOMES:
Cortical Blood Deoxygenation reactivity to hypercapnia using functional near-infrared spectroscopy (fNIRS) | Change from baseline to 2 hours
  Cerebral deoxygenated haemoglobin minimal levels in the frontal cortical regions of the brain during the 5% carbon-dioxide breathing challenge (average across minutes 3 and 4 of breathing challenge)
Inverse Efficiency scores in a Modified version of the Stroop Task | 2 hours post intervention
  The modified Stroop included task blocks (designated as Colour match; Word match; Stroop and Double Stroop) of increasing difficulty so that performance could be compared between simple and more demanding tasks. Reaction time and accuracy of choice were recorded to estimate inverse efficiency scores (in seconds). Higher 'inverse efficiency scores' reflect worse performance on the task, whilst lower scores reflects better performance.
Flow-mediated dilatation (FMD) of the brachial artery using ultrasound (expressed as % FMD: change in brachial diameter from baseline to peak dilation following 5 minutes of arterial occlusion).. | Change from baseline to 2 hours
  FMD of the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Rendeiro, PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport, Exercise & Rehabilitation Sciences, University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No